CLINICAL TRIAL: NCT05424848
Title: Evaluation of Femoral Cartilage Thickness Ultrasonographic Measurement in Parkinson's Disease
Brief Title: Femoral Cartilage Thickness in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2022.01.3
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease; Articular Cartilage Disorder; Ultrasonography
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: Inclusion Criteria
  1. Having Parkinson's
  2. 50-75 years old
  Exclusion criteria
  1. Limited cooperation
  2. The patient has moderate to severe dementia or mental retardation, which may cause limitations in examination, testing and treatment
  3. The patient's refusal to participate in the study
  4. Application of total joint prosthesis for the knee area
  5. Secondary osteoarthritis
  Interventions: Other: Ultasonographic measurement
- Control group: Healthy control group
  Interventions: Other: Ultasonographic measurement

INTERVENTIONS:
Other: Ultasonographic measurement — Ultrasonographic measurements of the patients will be evaluated by Dr. Merve Damla Korkmaz. Patients will be positioned in a semi-dark room with the knees fully flexed. Ultrasonographic measurements will be made to evaluate the femoral cartilage thickness of both knees, with images taken from the suprapatellar axillary position. Images of the intercondylar area, lateral and medial femoral condyles of the right and left knees will be taken and the measurements will be made from these areas, 3 measurements will be taken from each knee and the average of these measurements will be taken.

SUMMARY:
Parkinson's Disease (PD) is a chronic, progressive, degenerative movement disorder characterized by motor and non-motor findings, and the incidence increases with age.There are different methods for the evaluation of articular cartilage in PD. The aim of this study is to examine the effect of cartilage thickness evaluated by US on disease stage, motor functions, balance and fall risks in individuals with Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a chronic, progressive, degenerative movement disorder characterized by motor and non-motor findings, and the incidence increases with age. It is the second most common neurodegenerative disease after Alzheimer's. Although the incidence of PD increases with age, early onset can also be seen in genetic variants. The prevalence of PD is 1% at the age of 65 and reaches 5% at the age of 85 years. Although the onset of the disease is usually between the ages of 65-70, the diagnosis is made under the age of 40 in 5% of patients. Although the progression process of PH varies between individuals, it has physical, psychological and socioeconomic effects on patients and families in the later stages of the disease. In the advanced stages of the disease, serious complications can be seen, including pneumonia, which can cause mortality.During the course of the disease, rigidity, resting tremor, postural instability, gait disturbance and bradykinesia characterized by progressive decrease in speed and amplitude of repetitive movements are the main cardinal motor findings. In addition to these findings, secondary motor symptoms such as bradymymia, dysarthria, and associated movements in the arm accompany the disease during its course.There are different methods for the evaluation of articular cartilage. Although arthroscopy is the most reliable of these methods, the fact that it is an invasive method limits its applicability. Magnetic Resonance imaging, on the other hand, is a reliable and non-invasive method, but it is expensive and some patients do not prefer this method due to claustrophobia, which limits its use. Although the most commonly used method today is conventional radiography, this method is insufficient to evaluate cartilage thickness. In recent years, ultrasonography (US) has found a very wide area of use for physicians dealing with musculoskeletal diseases.US is accepted as a cost-effective method that allows the patient to feel the least discomfort, provides simultaneous imaging, and allows repeated dynamic evaluations.In addition to being used in the diagnosis and follow-up of various diseases, it allows quantitative measurements of various structures. Likewise, in vivo and in vitro studies have reported that sagittal and axial measurements of femoral cartilage thickness using US measurement are reliable. The most important disease associated with cartilage loss in the literature is osteoarthritis.

The aim of this study is to examine the effect of cartilage thickness evaluated by US on disease stage, motor functions, balance and fall risks in individuals with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Having Parkinson's
* 50-75 years old

Exclusion Criteria:

* Limited cooperation
* The patient has moderate to severe dementia or mental retardation, which may cause limitations in examination, testing and treatment
* The patient's refusal to participate in the study
* Application of total joint prosthesis for the knee area
* Secondary osteoarthritis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study sample will be included with Parkinson's Disease Patient and healthy control group.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic measurement | Baseline
  Images of the intercondylar area, lateral and medial femoral condyles of the right and left knees will be taken and the measurements will be made from these areas, 3 measurements will be taken from each knee and the average of these measurements will be taken.
The Hoehn and Yahr Scale | Baseline
  All patients in this study were classified based on the Hoehn and Yahr scale prior to treatment. This scale is widely used for classifying PD into five stages. It permits objective evaluation of the progression of the disease, from Stage 0 (no disease symptoms) to Stage 5 (the patient is confined to a wheelchair or bed)
The Movement Disorder Society Unified Parkinson's Disease rating Scale (MDS-UPDRS) | Baseline
  This is an extensive scale employed for the clinical evaluation of severity of PD. It consists of four sections including non-motor findings, motor problems, motor findings, and treatment complications

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Baseline
  The BDI is used to evaluate physical, emotional, and cognitive symptoms encountered in depression, such as hopelessness, irritability, guilt, fatigue, and weight loss. Scoring is performed from absence of symptoms to severe symptoms. Total scores range between 0 (no depression) and 63 (severe depression).
International Falls Efficacy Scale (FES) | Baseline
  This 10-question scale evaluated the individual's daily living activities. Subjects are asked how safe they feel when performing these activities, each question being scores from 1 (not at all concerned) to 10 (very concerned). Scoring is based out of a total possible score of 100, with scores of 70 or more indicating a fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: merve damla korkmaz, M.D., Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)